CLINICAL TRIAL: NCT04488536
Title: Management and Outcomes of Patients Admitted to Coronary Care Units, Depending on Degree of Frailty and Comorbidities
Status: Active, not recruiting | Type: Observational
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Niklas Ekerstad, Associate professor, Linkoeping University
Other Study IDs: 2020-01708
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Myocardial Infarction; Frailty
Keywords: Myocardial infarction; Frailty assessment; Clinical Frailty Scale; Predictive power; Mortality
MeSH Terms: conditions — Myocardial Infarction; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail patients: Clinical Frailty Scale level 5-9
  Interventions: Diagnostic Test: Clinical Frailty Scale
- Nonfrail patients: Clinical Frailty Scale level 1-4
  Interventions: Diagnostic Test: Clinical Frailty Scale

INTERVENTIONS:
Diagnostic Test: Clinical Frailty Scale — Frailty assessment

SUMMARY:
Background Patients less than 80 years of age, who suffer a myocardial infarction (MI) are usually (>90%) offered an early invasive strategy including coronary angiography possibly followed by intervention, preferably percutaneous coronary intervention (PCI). Among non ST-elevation myocardial infarction (NSTEMI) patients, 80 years of age or over, only approximately 40% receive an invasive approach in Sweden, since the majority are handled in a conservative way, i.e. with medical treatment only. Furthermore, as with pharmacological treatment, there is a large variation between Swedish counties regarding the choice of strategy for the treatment of elderly (80+) patients with NSTEMI with an even larger variation between acute hospitals ranging from 20% to 90 %.

The Swedish national guidelines for heart disease have emphasized that the patient's biological age, i.e. the patient's biological status and expected length of life, is crucial for decision-making. The Clinical Frailty Scale (CFS) is a global clinical measure of biological age, mixing co-morbidity, disability and cognitive impairment. The investigators have previously reported the potential importance of frailty for short-term (1 month) and medium-term outcome (1 year) in a NSTEMI population. However, published data on the role of frailty´s prognostic value, its capacity to predict adverse effects including complications, and the potential to guide clinical decision-making for elderly patients with myocardial infarction are scarce. Similarly, there is a lack of knowledge of how different patterns of comorbidity burden might influence rational decision-making.

Aims To explore the association between frailty and treatment patterns in cardiac care To study the association between outcomes and degree of frailty, with and without comprehensive adjustment for differences in baseline characteristics.

To study how treatment benefits for patients admitted to coronary care units differ in patients depending on comorbidities and frailty.

Hypothesis The investigators hypothesize that frailty is independently associated with worse outcomes, including mortality, readmissions and complications.

Methods and material An observational, register based, multicentre study. Inclusion criteria: Patients consecutively included in the Swedish Web-System for Enhancement and Development of Evidence-Based Care in Heart Disease Evaluated According to Recommended Therapies (SWEDEHEART) registry. Exclusion criteria: None.

SWEDEHEART is a national quality registry collecting information on all patients hospitalized with MI or suspected MI. All 72 Swedish hospitals with acute coronary care contribute with data. Briefly, information is collected prospectively about individual patients' medical history, treatment before admission, management during hospital stay, treatment at discharge, and diagnoses. Approximately 20.000 patients diagnosed with MI are included in this register per year. From January 1st 2020 frailty (CFS) is a mandatory variable in the registry. However, as a pilot project to ensure feasibility, five hospitals began to register frailty November 1st, 2017. For the investigators initial analyses data will be used from the pilot study to assess the association between CFS level and outcomes. The data extraction will be done by one of the monitors of the SWEDEHEART registry. After about two years the investigators will extract data prospectively entered into the registry.

The frailty instrument The crucial study instrument CFS is a 9-point scale. It has good predictive validity and prognostic power, is relying on clinical judgment, and is relatively easily used in clinical practice. Since the scale includes several degrees it can be considered to be particularly appropriate for risk stratification, and accordingly it has been used for this purpose. The investigators have got the instrument owner´s permission to use this scale.

The case record form (CRF) focus on demographic and clinical patient characteristics registered in the SWEDEHEART, particularly those which are supposed to be potential confounders when testing the hypothesis: chronological age, gender, cardiovascular risk, diabetes, heart failure, renal insufficiency, other co-morbidities, including the Charlson Comorbidity Index (CCI), previous MI, medications, ejection fraction, and the classification of MI. Cardiovascular risk will be assessed according to the Global Registry of Acute Coronary Events (GRACE) risk score (GRS). Results from echocardiography, ECGs, laboratory testing and registration of anthropometric data will be included according to routine practice within the frame of SWEDEHEART.

Follow-up of cohorts of invasively or conservatively treated patients with different stages of frailty will be done one, three, six, 12, 24 and 36 months after the inclusion point respectively.

DETAILED DESCRIPTION:
Background In Western countries the numbers of elderly patients are increasing. Although many elderly individuals are healthy, the number of individuals with complex needs for health care is large and growing. Patients less than 80 years of age, who suffer a myocardial infarction are usually offered an early invasive strategy including coronary angiography possibly followed by intervention, preferably percutaneous coronary intervention (PCI). Among non ST-elevation myocardial infarction (NSTEMI) patients, 80 years of age or over, only approximately 40% receive an invasive approach in Sweden, since the majority are handled in a conservative way, i.e. with medical treatment only. Furthermore, as with pharmacological treatment, there is a large variation between Swedish counties regarding the choice of strategy for the treatment of elderly (80+) patients with NSTEMI with an even larger variation between acute hospitals ranging from 20% to 90 %.

The Swedish national guidelines for heart disease have emphasized that the patient's biological age, i.e. the patient's biological status and expected length of life, is crucial for decision-making, though there is limited guidance regarding how the biological age should be estimated.The term frailty denotes a multi-dimensional syndrome characterized by increased vulnerability and decreased physiologic reserves, which can be seen as a marker of biological age.

The Canadian Study of Health and Ageing (CSHA) Clinical Frailty Scale (CFS) is a global clinical measure of biological age, mixing co-morbidity, disability and cognitive impairment. The CFS might be the most commonly used frailty instrument in an acute care context. The investigators have previously reported the potential importance of frailty for short-term (1 month) and medium-term outcome (1 year) in a NSTEMI population. However, published data on the role of frailty´s prognostic value, its capacity to predict adverse effects including complications, and the potential to guide clinical decision-making for elderly patients with myocardial infarction are scarce, particularly regarding longer-term outcomes.Similarly, there is a lack of knowledge of how different patterns of comorbidity burden, e.g. measured by a well-established index like the Charlson Comorbidity Index (CCI) might influence rational decision-making. Particularly this might be true regarding the combination of frailty and comorbidity.

The large variation in the management of these patients shows that there is need for further studies within this area in order to determine which treatment one should chose, whether it be invasive or conservative, in different groups.

Aims To explore the association between frailty and treatment patterns in cardiac care To study the association between outcomes and degree of frailty, with and without comprehensive adjustment for differences in baseline characteristics.

To study how treatment benefits for patients admitted to coronary care units differ in patients depending on comorbidities and frailty.

Hypothesis The investigators hypothesize that frailty is independently associated with worse outcomes, including mortality, readmissions and complications.

The investigators also hypothesize that frailty influences the benefit-risk ratio for pharmacological therapies and invasive treatments.

Methods and material An observational, register based, multicentre study. Inclusion criteria: Patients consecutively included in the SWEDEHEART registry. Exclusion criteria: None.

SWEDEHEART is a national quality registry collecting information on all patients hospitalized with MI or suspected MI. All 72 Swedish hospitals with acute coronary care contribute with data. Briefly, information is collected prospectively about individual patients' medical history, treatment before admission, management during hospital stay, treatment at discharge, and diagnoses. Approximately 20.000 patients diagnosed with MI are included in this register per year. From January 1st 2020 frailty (CFS) is a mandatory variable in the registry. However, as a pilot project to ensure feasibility, five hospitals began to register frailty November 1st, 2017. These include three university hospitals: the Huddinge-Karolinska Hospital, the Linköping University Hospital and the Sahlgrenska Hospital, and two large county hospitals: The NAL-Uddevalla (NU) Hospital and Gavle Hospital. For the investigators initial analyses data will be used from the pilot study to assess the association between CFS level and outcomes. The data extraction will be done by one of the monitors of the SWEDEHEART registry. After about two years the investigators will extract data prospectively entered into the registry. By use of the Swedish unique personal identification numbers (PIN) data from the SWEDEHAERT will be merged with data from the National cause of death registry in order to obtain information on mortality and cause of death, with the National patient registry, a comprehensive national register of the consumption of inpatient hospital care maintained by the Swedish National Board of Health and Welfare, to obtain information on comorbidity and outcomes, with the Swedish prescribed drugs registry to obtain information on collected drugs and from Statistics Sweden information on socio-economic factors and country of birth. After data extraction, merging PINs will be removed and all statistical analyses will be performed on de-identified data.

The frailty instrument The crucial study instrument CFS is a 9-point scale, derived from the deficit of accumulation model of frailty, and it has been validated against the Frailty Index. It has good predictive validity and prognostic power, is relying on clinical judgment, and is relatively easily used in clinical practice, see the attached document Clinical Frailty Scale. Since the scale includes several degrees it can be considered to be particularly appropriate for risk stratification, and accordingly it has been used for this purpose. The investigators have got the instrument owner´s permission to use this scale.

The evaluation of the patient's degree of frailty will be based on bedside judgment undertaken preferably by registered nurses regarding frailty and other clinical information including the records in the patient file. The inter-rater reliability among a sample of frailty-assessing nurses will be pragmatically assessed before the study start, see Statistics. During the study there will be several support functions in order to enhance the validity and reliability of the judgments: a manual and an instruction film on the frailty assessment via CFS has been developed by a focus group including cardiological and geriatric expertise; there will be instructions on how to assess frailty on the homepage of SWEDEHEART; and five trained SWEDEHEART nurses will function as monitors and support for the local assessing nurses, as will the mentioned expert group.

The CRF focus on demographic and clinical patient characteristics registered in the SWEDEHEART, particularly those which are supposed to be potential confounders when testing the hypothesis: chronological age, gender, cardiovascular risk, diabetes, heart failure, renal insufficiency, other co-morbidities, including the Charlson Comorbidity Index (CCI), previous MI, medications, ejection fraction, and the classification of MI. Cardiovascular risk will be assessed according to the Global Registry of Acute Coronary Events (GRACE) risk score (GRS).

Results from echocardiography, ECGs, laboratory testing and registration of anthropometric data will be included according to routine practice within the frame of SWEDEHEART.

Follow-up of cohorts of invasively or conservatively treated patients with different stages of frailty will be done one, three, six, 12, 24 and 36 months after the inclusion point respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively included in the SWEDEHEART registry from November 1, 2017.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: SWEDEHEART is a national quality registry, which collects information on all patients hospitalized with MI or suspected MI. All 72 Swedish hospitals with acute coronary care contribute with data. From January 1st 2020 Clinical Frailty Scale, the 9-degree-version (CFS-9) is a mandatory variable in the registry. However, as a pilot project to ensure feasibility, five hospitals began to register frailty November 1st, 2017. Inclusion criteria: patients consecutively included in the SWEDEHEART registry from November 1, 2017. Exklusion criteria: none.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Mortality rate by 6 months after inclusion. | 6 months after inclusion
  Mortality rate (death from any cause) by 6 months after inclusion.

SECONDARY OUTCOMES:
Mortality rates up to 36 months after inclusion. | 3-36 months after inclusion
  Mortality rates (death from any cause) up to 36 months after inclusion (measured at 3, 12, 24, 36 months)
Rates of readmissions and complications up to 36 months after inclusion. | 3-36 months after inclusion
  Rates of readmissions, re-infarctions, major bleedings and other complications up to 36 months after inclusion (measured at 3, 12, 24, 36 months)
Description of treatment patterns including medications and invasive strategies from admission to hospital (inclusion) to discharge from hospital (index care hospital episode) | From admission to hospital (inclusion) up to 36 months after inclusion
  Percentage (%) of patients receiving evidence based medications during the index care hospital episode Percentage (%) of patients receiving evidence based interventions during the index care hospital episode

CONTACTS AND LOCATIONS:
Overall Officials: Niklas Ekerstad, MD, PhD, Principal Investigator — Linkoeping University
Locations (2):
- Sweden (2):
  - Linkoeping University Hospital, Linköping, Ostergoetland
  - The Center for Medical Technology Assessment/IMH, Linkoeping University, Linköping, Östergötland County

IPD SHARING:
Plan to Share IPD: No